CLINICAL TRIAL: NCT07232368
Title: The Effect of Slow-Paced Breathing on Patient Outcomes in Pulmonary Arterial Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Fikriye Ersel, lecturer, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 22-AKD-202
Record Dates: First submitted 2025-11-13; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Arterial Hypertension (PAH) (WHO Group 1 PH)
Keywords: Pulmonary Arterial Hypertension; Slow-paced Breathing; Symptom Management; Quality of life; Nursing
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Intervention Model Description: It consists of two groups, application and control
Who Masked: Participant, Outcomes Assessor
Masking Description: In this randomized controlled experimental study, Excel random numbers function was used as the randomization method.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Data collection tools were applied to individuals in the control group at week 0 (first follow-up), week 6 (interim follow-up) and week 12 (final follow-up) of the follow-up period.
  The data collection tools administered to the control group were: Patient Identification Form, Multidimensional Dyspnea Profile, Multidimensional Fatigue Inventory, Pittsburgh Sleep Quality Index, Six-Minute Walk Test Form and Modified Borg Scale, Laboratory Analysis Form, and EmPHasis-10 Quality of Life Scale, Digital Literacy Scale-Technical Subscale.
- initiative group (Experimental): Data collection tools were administered to individuals in the intervention group at week 0 (initial follow-up), week 6 (interim follow-up), and week 12 (final follow-up).
  Data collection tools administered to the intervention group included:
  Patient Identification Form, Multidimensional Dyspnea Profile, Multidimensional Fatigue Inventory, Pitsburgh Sleep Quality Index, Six-Minute Walk Test Form and Modified Borg Scale, Laboratory Analysis Form, EmPHasis-10 Quality of Life Scale, Digital Literacy Scale-Technical Subscale.
  Interventions: Other: Slow-paced breathing intervention

INTERVENTIONS:
Other: Slow-paced breathing intervention — Other: Slow-paced breathing intervention After the intervention and control groups were determined, the purpose of the study was explained to both groups. Participants were informed that the intervention would last 12 weeks. Data collection forms would be completed face-to-face before the intervention (initial follow-up), during the 6th week (interim follow-up), and at the 12th week (final follow-up).
  Patients in the intervention group received a slow-paced breathing intervention in addition to the standard treatment protocol (verbal, video, and hands-on instruction, demonstration). After the first interview, participants received the application video (installed on a device such as a mobile phone, personal computer, and/or tablet, depending on the participant's preference and ease of use).
  The control group received only the standard treatment protocol. However, they were informed that they could perform the slow-paced breathing intervention upon completion of the study if they wished
  Arms: initiative group

SUMMARY:
This study aims to investigate the effects of slow-paced breathing (SPB) intervention applied to patients with pulmonary arterial hypertension (PAH) in the home environment on symptom management (dyspnea, fatigue, sleep quality), clinical parameters (Six-Minute Walking Test-6MWT), IL-6, NT-proBNP results) and quality of life.

DETAILED DESCRIPTION:
The therapeutic power of slow, controlled breathing has been recognized for centuries and is primarily used in relaxation techniques such as meditation and yoga.

It can be difficult for a patient to effectively perform these exercises on their own without training or individualized coaching.

Numerous studies in recent years have shown that therapeutic breathing exercises performed without conscious effort, using devices, have positive effects on parameters such as blood pressure, stress management, respiratory modulation, sleep difficulties, and quality of life.

Furthermore, the effects of slow-paced breathing performed with conscious effort using visual and auditory triggers have also been demonstrated in many studies.

Slow-paced breathing is a breathing technique that aims to slow the inhalation and exhalation phases to a controlled rate determined by a visual, auditory, or kinesthetic pacer.

While the spontaneous respiratory rate in adults is generally between 12 and 20 breaths per minute, this rate is reduced to as little as 6 breaths per minute with slow-paced breathing.

With the therapeutic use of slow-paced breathing intervention, Studies have shown that arterial baroreflex sensitivity is increased, cardiopulmonary reflexes are activated, vascular resistance is reduced, peripheral blood flow is increased, and many positive effects on the cardiovascular system and respiratory functions, including respiratory sinus arrhythmia and exercise tolerance.

There are very few studies on the outcomes of interventions aimed at symptom control, one of the most important goals of nursing care in pulmonary arterial hypertension.

The existing studies (only two) are foreign-based and uncontrolled experimental studies. While they demonstrate the positive effects of the interventions, they cannot provide comprehensive data and have limited evidence. Further studies are needed to provide sufficient evidence on the subject. Furthermore, a systematic review of the existing literature revealed that studies on PAH, a rare disease, are quite limited at all levels. The nursing literature is even more limited.

A video of a slow-paced breathing practice was used as an educational material in our research.

This video was prepared with expert support based on videos used in similar studies for educational and demonstration purposes.

The video preparation process: The presentation began with the preparation of a PowerPoint presentation using Microsoft Office 365 on a computer. The PowerPoint program's video conversion feature was used to make the presentation accessible on all platforms (Windows, iOS, Android, etc.).

The video included a visual guide (a moving ball) that was followed visually to ensure adherence to a predetermined breathing rate, accompanied by relaxing music. This visual guide asked patients to continuously inhale through the nose as the ball rose, and to continuously exhale through the mouth with pursed lips as the ball descended.

This study, which investigates the effects of slow-paced breathing intervention applied at home in patients with pulmonary arterial hypertension on symptom management, clinical parameters, and quality of life, is a study that will contribute to the literature on cardiology nursing in our country and around the world.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 65 years of age
* Being diagnosed with PAH (pulmonary arterial hypertension)- (Group I pulmonary hypertension (idiopathic, hereditary, drug or toxin-induced, or associated with connective tissue disease, congenital heart disease, or HIV-associated)) diagnosed by right heart catheterization
* Being on stable PAH treatment for the past three months and in a stable clinical condition (no changes in PAH medical treatment, no new medications added)
* Being in class II or III according to the World Health Organization functional classification
* Being able to speak Turkish
* Having a high level of technical digital literacy (obtaining the highest score (30 points) on the "technical subscale" of the Digital Literacy Scale*)
* Agreeing to participate in the study

Exclusion Criteria:

* Communication difficulties
* Symptomatic hypotension
* Pregnancy status for female participants (positive urine pregnancy test*)
* Presence of another underlying condition that may cause dyspnea, fatigue, and sleep difficulties (chronic fatigue syndrome, obstructive sleep apnea, restless legs syndrome, narcolepsy, major depression, etc.)
* Hospitalization or acute phase
* Active participation in a cardiac rehabilitation program
* Presence of pulmonary hypertension due to left heart disease and pulmonary hypertension due to lung diseases and/or hypoxia
* Receiving a lung transplant
* Having had cardiac surgery within the last six months
* Presence of obesity
* Presence of mental retardation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-06-11 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Multidimensional Dyspnea Profile | Baseline, at the end of six weeks and at the end of twelve weeks
  The multidimensional dyspnea profile consists of subheadings assessing immediate perception (6 items; total score range 0-60) and emotional reactions (5 items; total score range 0-50). Items are rated on a 0-10 scale, with higher scores indicating greater intensity, unpleasantness, or distress.
Multidimensional Fatigue Inventory | Baseline, at the end of six weeks and at the end of twelve weeks
  The inventory contains five subscales measuring general fatigue (items 1, 5, 12, and 16), physical fatigue (items 2, 8, 14, and 20), decreased activity (items 3, 6, 10, and 17), decreased motivation (items 4, 9, 15, and 18), and mental fatigue (items 7, 11, 13, and 19), totaling 20 items.
Pittsburgh Sleep Quality Index | Baseline, at the end of six weeks and at the end of twelve weeks
  The index is a self-report measure that provides a quantitative measure of sleep quality to describe good and poor sleep over a one-month period. It consists of seven subcomponents and 24 items, 19 of which are self-reported and five of which are self-reported or evaluated by a roommate, if present.
Six-Minute Walk Test Form and Modified Borg Scale | Baseline, and at the end of twelve weeks
  The 6MWT (Six-Minute Walk Test), the most commonly used exercise test in monitoring patients with pulmonary hypertension, is an easy-to-administer and inexpensive test. Walking speed should be determined by the patient, but the goal of the test is to walk as far as possible in six minutes.
  The Modified Borg Scale, a unidimensional scale, is a subjective, reliable, and easily administered tool for determining the severity of dyspnea and fatigue perceived by the patient at rest and during exertion. The scale identifies the severity of dyspnea/fatigue by rating (0 to 10), with a score of 0 indicating "absent" and a score of 10 indicating "maximum" dyspnea/fatigue.
Laboratory Analysis Form | Baseline, and at the end of twelve weeks
  It is recommended to monitor certain variables (NT-proBNP) at regular intervals during the diagnosis and follow-up phases of the disease. These variables can be used to assess prognosis and risk stratify, while also guiding the treatment protocol.
  In addition, some studies have used IL-6 as an indicator of inflammation and correlated it with sleep quality.
EmPHasis-10 Quality of Life Scale | Baseline, at the end of six weeks and at the end of twelve weeks
  This 10-question scale, developed for patients with pulmonary hypertension, addresses concerns about the disease's significant effects, such as shortness of breath, fatigue, and lack of energy, as well as its impact on social relationships. Each question on the scale has a score between 0 and 5 and is assessed using a Likert scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege Üniversitesi, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No